CLINICAL TRIAL: NCT00230061
Title: Randomised Open Label Clinical Trial of the Immune Response to Hepatitis B Vaccination in HIV-infected Persons.
Brief Title: Hepatitis B Vaccination in HIV-infected Persons
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Collaborators: Stichting Nuts Ohra (Other)
Responsible Party: Theodora EMS de Vries-Sluijs, ErasmusMC
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SNO-T-07-102
Record Dates: First submitted 2005-09-28; First posted 2005-09-30 (Estimated); Last update posted 2010-06-02 (Estimated); Status verified 2010-06

CONDITIONS: HIV Infections; Hepatitis B
Keywords: HIV
MeSH Terms: conditions — HIV Infections; Hepatitis B | interventions — Hepatitis B Vaccines; Vaccines

INTERVENTIONS:
Biological: HBVAXPRO, Hepatitis B (Recombinant) vaccine, 10 mcg/ml

SUMMARY:
In this study we compare the efficacy of two different HBV-vaccination schedules in HIV-infected persons concerning immune response and compliance. Short schedule: t=0,1,3 weeks and standard schedule: t=0,1,6 months.

DETAILED DESCRIPTION:
It is known that HIV-infected persons are more prone to develop chronic hepatitis B infection when they get infected with this virus. After developing chronic hepatitis B these patients are more likely to get livercirrosis and hepatocellular carcinoma (Bodsworth et al.).

Hepatitis B vaccination is available and the vaccine is about 95% protective in preventing immunocompetent persons from developing chronic hepatitis B infection (Lemon). The response on this vaccin is less effective in HIV-infected persons (Carne et al.). Furthermore there is a compliance problem in the standard scheme.

In this study we compare the efficacy of two different HBV vaccination schedules in HIV-infected persons concerning immune response and compliance. A short schedule: t=0,1,3 weeks, in which there are good results concerning immune response and compliance in immunocompetent persons (Saltog et al.) and the standard schedule: t=0,1,6 months. Patients not immune at week 28 will be offered boostervaccination. This consists of double doses at t=0,1,2 months.

800 persons are needed to show non-inferiority with lower margin of 10% of the short schedule in comparison with the control group. Powercalculation is 80%. Randomization is stratified according to CD4 count(CD4 <200, 200-500, >500).

The hypothesis of the study is a better compliance and a comparable immune response in the short schedule, through which persons will be protected against hepatitis B in an early stage.

ELIGIBILITY:
Inclusion Criteria:

* HIV positive
* Negative for HBsAg and anti-HBc
* 18 years or older

Exclusion Criteria:

* previous Hepatitis B vaccination
* current opportunistic infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2004-04; Primary Completion 2008-05 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Measurement of anti-Hbs titer after completing hepatitis B vaccination.

SECONDARY OUTCOMES:
To compare response and compliance between two vaccination schedules: short and standard

CONTACTS AND LOCATIONS:
Overall Officials: Theodora EM de Vries-Sluijs, MD, Principal Investigator — Erasmus Medical Center
Locations (1):
- Erasmus Medical Center, Rotterdam, Netherlands

REFERENCES:
- [Background] Bodsworth NJ, Cooper DA, Donovan B. The influence of human immunodeficiency virus type 1 infection on the development of the hepatitis B virus carrier state. J Infect Dis. 1991 May;163(5):1138-40. doi: 10.1093/infdis/163.5.1138. PMID 2019762
- [Background] Sinicco A, Raiteri R, Sciandra M, Bertone C, Lingua A, Salassa B, Gioannini P. Coinfection and superinfection of hepatitis B virus in patients infected with human immunodeficiency virus: no evidence of faster progression to AIDS. Scand J Infect Dis. 1997;29(2):111-5. doi: 10.3109/00365549709035869. PMID 9181644
- [Background] Ockenga J, Tillmann HL, Trautwein C, Stoll M, Manns MP, Schmidt RE. Hepatitis B and C in HIV-infected patients. Prevalence and prognostic value. J Hepatol. 1997 Jul;27(1):18-24. doi: 10.1016/s0168-8278(97)80274-7. PMID 9252068
- [Background] Lemon SM, Thomas DL. Vaccines to prevent viral hepatitis. N Engl J Med. 1997 Jan 16;336(3):196-204. doi: 10.1056/NEJM199701163360307. No abstract available. PMID 8988900
- [Background] Carne CA, Weller IV, Waite J, Briggs M, Pearce F, Adler MW, Tedder RS. Impaired responsiveness of homosexual men with HIV antibodies to plasma derived hepatitis B vaccine. Br Med J (Clin Res Ed). 1987 Apr 4;294(6576):866-8. doi: 10.1136/bmj.294.6576.866. PMID 3105779
- [Background] Keet IP, van Doornum G, Safary A, Coutinho RA. Insufficient response to hepatitis B vaccination in HIV-positive homosexual men. AIDS. 1992 May;6(5):509-10. No abstract available. PMID 1535502
- [Background] Wong EK, Bodsworth NJ, Slade MA, Mulhall BP, Donovan B. Response to hepatitis B vaccination in a primary care setting: influence of HIV infection, CD4+ lymphocyte count and vaccination schedule. Int J STD AIDS. 1996 Nov-Dec;7(7):490-4. doi: 10.1258/0956462961918563. PMID 9116065
- [Background] Bruguera M, Cremades M, Salinas R, Costa J, Grau M, Sans J. Impaired response to recombinant hepatitis B vaccine in HIV-infected persons. J Clin Gastroenterol. 1992 Jan;14(1):27-30. doi: 10.1097/00004836-199201000-00007. PMID 1532609
- [Background] Rey D, Krantz V, Partisani M, Schmitt MP, Meyer P, Libbrecht E, Wendling MJ, Vetter D, Nicolle M, Kempf-Durepaire G, Lang JM. Increasing the number of hepatitis B vaccine injections augments anti-HBs response rate in HIV-infected patients. Effects on HIV-1 viral load. Vaccine. 2000 Jan 18;18(13):1161-5. doi: 10.1016/s0264-410x(99)00389-8. PMID 10649616
- [Background] Sasaki Md, Foccacia R, de Messias-Reason IJ. Efficacy of granulocyte-macrophage colony-stimulating factor (GM-CSF) as a vaccine adjuvant for hepatitis B virus in patients with HIV infection. Vaccine. 2003 Nov 7;21(31):4545-9. doi: 10.1016/s0264-410x(03)00500-0. PMID 14575766
- [Background] Wilson CM, Ellenberg JH, Sawyer MK, Belzer M, Crowley-Nowick PA, Puga A, Futterman DC, Peralta L; Adolescent Medicine HIV/AIDS Research Network. Serologic response to hepatitis B vaccine in HIV infected and high-risk HIV uninfected adolescents in the REACH cohort. Reaching for Excellence in Adolescent Care and Health. J Adolesc Health. 2001 Sep;29(3 Suppl):123-9. doi: 10.1016/s1054-139x(01)00278-6. PMID 11530313
- [Background] Rutstein RM, Rudy B, Codispoti C, Watson B. Response to hepatitis B immunization by infants exposed to HIV. AIDS. 1994 Sep;8(9):1281-4. doi: 10.1097/00002030-199409000-00010. PMID 7802981
- [Background] Scolfaro C, Fiammengo P, Balbo L, Madon E, Tovo PA. Hepatitis B vaccination in HIV-1-infected children: double efficacy doubling the paediatric dose. AIDS. 1996 Sep;10(10):1169-70. No abstract available. PMID 8874636
- [Background] Saltoglu N, Inal AS, Tasova Y, Kandemir O. Comparison of the accelerated and classic vaccination schedules against Hepatitis B: three-week Hepatitis B vaccination schedule provides immediate and protective immunity. Ann Clin Microbiol Antimicrob. 2003 Nov 17;2:10. doi: 10.1186/1476-0711-2-10. PMID 14622443
- [Background] Marchou B, Picot N, Chavanet P, Auvergnat JC, Armengaud M, Devilliers P, Cerisier JE, Marie FN, Excler JL. Three-week hepatitis B vaccination provides protective immunity. Vaccine. 1993 Nov;11(14):1383-5. doi: 10.1016/0264-410x(93)90165-t. PMID 8310757
- [Background] Nothdurft HD, Dietrich M, Zuckerman JN, Knobloch J, Kern P, Vollmar J, Sanger R. A new accelerated vaccination schedule for rapid protection against hepatitis A and B. Vaccine. 2002 Jan 15;20(7-8):1157-62. doi: 10.1016/s0264-410x(01)00432-7. PMID 11803077
- [Background] Wright NM, Campbell TL, Tompkins CN. Comparison of conventional and accelerated hepatitis B immunisation schedules for homeless drug users. Commun Dis Public Health. 2002 Dec;5(4):324-6. PMID 12564251